CLINICAL TRIAL: NCT05448976
Title: Potential Effect for the Smoking on Periodontitis From the Perspective of Arginine Metabolites Symmetric Dimethylarginine (SDMA) and Asymmetric Dimethylarginine (ADMA)
Brief Title: Potential Effect for the Smoking on Periodontitis From the Perspective of Arginine Metabolites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Nur Balci, DDs, PhD, ASSOC. PROF DR, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 781
Record Dates: First submitted 2022-06-29; First posted 2022-07-08 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2022-07

CONDITIONS: Periodontitis; Smoking; Inflammatory Response
Keywords: Periodontitis, Arginine metabolites, Smoking
MeSH Terms: conditions — Periodontitis; Smoking

STUDY DESIGN:
Intervention Model Description: Saliva and serum of periodontitis and smoking patients collected for analyzing arginine metabolites.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saliva and serum collection of patients and samples molecules analysis (Active Comparator): aliva and serum sampling Saliva were collected to analyze the selected markers as unstimulated samples during the early hours of the day. The saliva was centrifuged and then transferred into Eppendorf tubes. Venous puncture was performed after saliva collection and 10 mL of blood samples were collected by qualified staff (MY,EY) from each participant. Saliva and serum were then stored at -80 °C until analysis.
  Interventions: Other: Saliva and serum sampling
- Salivary and serum arginine metabolites ADMA and SDMA observation (Experimental): IL-6 levels in collected samples were determined by ELISA kits and analyzed according to manufacturers' instructions, with colorimetric assessment performed using a microplate reader at 450 nm with the assay detection range between 7.8 and 500 pg/mL. Concentrations were determined based on the respective assay standard curve. All samples were analyzed in duplicate, and the average was used in subsequent calculations.
  Determination of methylated arginine metabolites:
  The ADMA, SDMA, homoArg, arginine and L-NMMA levels in saliva and serum were assessed by a liquid chromatography-mass spectrometry (LC MS/MS)* method, which was a modification of the method of Di Gangi et al.
  Interventions: Other: Saliva and serum sampling

INTERVENTIONS:
Other: Saliva and serum sampling — Saliva were collected to analyze the selected markers as unstimulated samples during the early hours of the day. The saliva was centrifuged and then transferred into Eppendorf tubes. Venous puncture was performed after saliva collection and 10 mL of blood samples were collected by qualified staff (MFD) from each participant. Saliva and serum were then stored at -80 °C until analysis.

SUMMARY:
Arginine metabolites are amino acids that are associated with vascular tone regulation and the level of inflammation, with critical roles in the synthesis of NO. Our aim was to determine the ADMA, SDMA, L-NMMA, L-arginine, L-homoarginine and IL-6 levels in saliva and serum samples from periodontitis patients and periodontally healthy individuals and to assess the levels of these compounds according to smoking status and compare these levels to those of healthy individuals.

DETAILED DESCRIPTION:
The study consisted of four groups: healthy individuals (control (C); n=20), smokers with healthy periodontium (S-C; n=20), nonsmokers with Stage III Grade B generalized periodontitis (P; n=20) and smokers with Stage III Grade C generalized periodontitis (S-P; n=18). Clinical periodontal parameters were measured. The determination of methylated arginine metabolites was carried out by LC-MS/MS.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy
* clinical diagnosis of periodontitis
* clinical diagnosis of periodontal health
* For smoking group the so kerr were denied as smoking at least 10 cigarettes per day and the duration should more than 10 years.

Exclusion Criteria:

* history of regular use of systemic antibiotics anti-inflammatory, or antioxidant drugs (previous 3 months)
* nonsurgical periodontal treatment (previous 6 months)
* surgical periodontal treatment (previous 12 months)
* presence of<10 teeth
* current medications affecting gingival health (calcium channel blockers, phenytoin, cyclosporine, and hormone replacement therapy)
* diabetes
* diagnosis of rheumatoid arthritis
* pregnancy
* lactating
* excessive alcohol consumption.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Pocket probing depth | 6 months
  Measurement of the depth of a sulcus or periodontal pocket determined by measuring distance from a gingival margin to the base of the sulcus or pocket with a calibrated periodontal probe
Clinical attachment level | 9 months
  Clinical attachment level (or loss, CAL) is a more accurate indicator of the periodontal support around a tooth than probing depth alone. CAL is measured from a fixed point on the tooth that does not change, the CEJ.
  To calculate CAL, two measurements are needed: distance from the gingival margin to the CEJ and probing depth.
  In recession: probing depth (+) gingival margin to the CEJ (add). In tissue overgrowth: probing depth (-) gingival margin to the CEJ (subtract)
Bleeding on probing | 9 months
  referring to bleeding that is induced by gentle manipulation of the tissue at the depth of the gingival sulcus, or interface between the gingiva and a tooth

SECONDARY OUTCOMES:
Saliva and serum samples processing | 2 months
  Phenomenex (Torrance, CA, USA) 75 x 4.6 mm x 4 µm polar-RP column, Dionex HPLC and Access MAX LC-MSMS (Thermo Scientific, USA) device were used; in the gradient phase mobile phase A (40 mM ammoniumformate, 3% formic acid) and mobile phase B (acetonitrile) were utilized. A flow chart with increasing in steps of 2-8 minutes for 10% B phase, 30% B phase for 8-11 minutes, and finally 10% B phase for 11-20 minutes was applied at a flow rate of 0.3 ml/min. MRM and CE values were as follows: Arginine 231.3-70.1 CE: 15 V; Homoarginine 245.2-84.2 CE: 24 V; L-NMMA 245.3-70.2 CE:15V; ADMA 259.3-214.0; CE:25V; SDMA 259.3-228.0 CE:15V; ADMA-D7 266.610-221.000 CE:15V; capillary temperature 210 °C; Vaporizer temperature 350 °C; Sheath gas pressure: 30 Arb.; Aux Gas pressure:10 Arb.; Ion Sweep Gas Pressure: 0; Spray Voltage: 3000 V; Polarity: (+).
serum and saliva analyses for arginine metabolites | 2 months
  The ADMA, SDMA, homoArg, arginine and L-NMMA levels in saliva and serum were assessed by a liquid chromatography-mass spectrometry (LC MS/MS)* method, which was a modification of the method of Di Gangi et al.

CONTACTS AND LOCATIONS:
Overall Officials: Nur Balci, Assoc Prof, Study Chair — Istanbul Medipol University.Istanbul Medipol University, School of Dentistry Istanbul, Fatih, Turkey, 34083
Locations (1):
- Istanbul Medipol University, School of Dentistry, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Di Gangi IM, Chiandetti L, Gucciardi A, Moret V, Naturale M, Giordano G. Simultaneous quantitative determination of N(G),N(G)-dimethyl-L-arginine or asymmetric dimethylarginine and related pathway's metabolites in biological fluids by ultrahigh-performance liquid chromatography/electrospray ionization-tandem mass spectrometry. Anal Chim Acta. 2010 Sep 16;677(2):140-8. doi: 10.1016/j.aca.2010.08.011. Epub 2010 Aug 17. PMID 20837180
- [Background] Tonetti MS, Greenwell H, Kornman KS. Staging and grading of periodontitis: Framework and proposal of a new classification and case definition. J Periodontol. 2018 Jun;89 Suppl 1:S159-S172. doi: 10.1002/JPER.18-0006. PMID 29926952
- [Background] Balci N, Kurgan S, Cekici A, Cakir T, Serdar MA. Free amino acid composition of saliva in patients with healthy periodontium and periodontitis. Clin Oral Investig. 2021 Jun;25(6):4175-4183. doi: 10.1007/s00784-021-03977-7. Epub 2021 May 11. PMID 33977387